CLINICAL TRIAL: NCT03984032
Title: Comparison of Clinical Performance of LMA Protector Cuff Pilot and LMA Supreme Among Anaesthetised, Non-Paralysed Patients
Brief Title: LMA Protector Cuff Pilot vs LMA Supreme Among Anaesthetised, Non-Paralysed Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liu Chian Yong (Other)
Responsible Party: Sponsor-Investigator, Liu Chian Yong, Consultant Anaesthesiologist, Universiti Kebangsaan Malaysia Medical Centre
Organization: Universiti Kebangsaan Malaysia Medical Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: UKM PPI/111/8/JEP-2018-007
Record Dates: First submitted 2019-05-16; First posted 2019-06-12 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Anesthesia
Keywords: LMA Protector Cuff Pilot; LMA Supreme; Clinical Performance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LMA Protector Cuff Pilot (Experimental)
  Interventions: Device: LMA Supreme
- LMA Supreme (Active Comparator)
  Interventions: Device: LMA Protector Cuff Pilot

INTERVENTIONS:
Device: LMA Protector Cuff Pilot — Assessing the clinical performance of LMA Protector Cuff Pilot
  Arms: LMA Supreme
Device: LMA Supreme — Assessing the clinical performance of LMA Supreme
  Arms: LMA Protector Cuff Pilot

SUMMARY:
Comparison of clinical performance between LMA Protector Cuff Pilot and LMA Supreme in terms of oropharyngeal leak pressure, time to insertion, ease of gastric tube insertion, laryngeal view, incidence of sore throat

ELIGIBILITY:
Inclusion Criteria:

* Patients planned for general anaesthesia without muscle relaxant usage via supraglottic airway device.

Exclusion Criteria:

* BMI > 35
* Patients with likelihood of difficult intubation (Simplified Airway Risk Index Score of 4 or more)
* Patients with increased risks of aspirations (gastrooesophageal reflux disease, obstetric patients, hiatus hernia)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2019-02-19 (Actual); Study Completion 2019-02-19 (Actual)

PRIMARY OUTCOMES:
Oropharyngeal leak pressure (OLP) | During induction of anaesthesia
  To assess the OLP of LMA Protector Cuff Pilot and LMA Supreme

SECONDARY OUTCOMES:
Mean time to insertion | During induction of anaesthesia
  To compare mean time to insertion of LMA Protector Cuff Pilot and LMA Supreme
Gastric tube insertion | After induction of anaesthesia
  To compare the ease of gastric tube insertion in LMA Protector Cuff Pilot and LMA Supreme
Laryngeal view | After induction of anaesthesia
  To compare the laryngeal view between LMA Protector Cuff Pilot and LMA Supreme
Complications | 24 hours
  To compare the incidence of sore throat and hoarseness of voice after insertion of LMA Protector Cuff Pilot and LMA Supreme

CONTACTS AND LOCATIONS:
Locations (1):
- Universiti Kebangsaan Malaysia Medical Centre, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Informed Consent Form (2018-07-14): https://cdn.clinicaltrials.gov/large-docs/32/NCT03984032/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2018-07-14): https://cdn.clinicaltrials.gov/large-docs/32/NCT03984032/Prot_SAP_001.pdf